CLINICAL TRIAL: NCT01776398
Title: Collection of Airway, Blood and/or Urine Specimens From Subjects for Research Studies
Status: Recruiting | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Boehringer Ingelheim (Industry); Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 1204012331; 1R01HL107882-01 (NIH)
Record Dates: First submitted 2012-10-10; First posted 2013-01-28 (Estimated); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Smoking; Smoking Cessation; Idiopathic Pulmonary Fibrosis (IPF); Rheumatoid Arthritis-Associated Interstitial Lung Disease; Scleroderma-Associated Interstitial Lung Disease (SSC-ILD)
Keywords: COPD; Chronic Obstructive Pulmonary Disease; Lung disease; Emphysema; Smoking; Healthy Smoker; Smoker; Non-smoker; IPF; RA-ILD; SSC-ILD; Idiopathic Pulmonary Fibrosis; Rheumatoid Arthritis-Associated Interstitial Lung Disease; Scleroderma-Associated Interstitial Lung Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Smoking; Smoking Cessation; Idiopathic Pulmonary Fibrosis; Lung Diseases; Emphysema

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Specimens collected may include blood, urine and airway samples (nasal, airway brushing, biopsy and/or washings) from consenting subjects. Subjects will include both individuals diagnosed with lung disease and healthy control subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 1.1 HEALTHY SUBJECTS: Healthy as defined by those not having lung disease and inclusive of: all races, ethnicities, sex, HIV status, smoking status and multiple birth status, etc., within the general population.
- 1.2 SUBJECTS WITH LUNG DISEASE: Defined by those having lung disease or symptoms of lung disease and inclusive of: all races, ethnicities, sex, HIV status, smoking status and multiple birth status, etc., within the general population)
- 2. WCMC/NYPH CLINICAL PATIENTS: Subjects may be recruited if subjects fit inclusion/exclusion criteria and are deemed eligible to participate as long as informed consent is given. Sample collection will occur during a separate study visit.
  WCMC/NYPH clinical patients will not undergo any additional procedures listed in this protocol as part of this research study.
- 3. PCNY CLINICAL PATIENTS: Subjects may be recruited if subjects fit inclusion/exclusion criteria and are deemed eligible to participate as long as informed consent is given. Sample collection will occur during a separate study visit. Clinical patients seen at the Pulmonary Consultants of New York will only undergo the nasal sample collection and may be asked to have a blood draw of about 2 teaspoons (9ml).

SUMMARY:
The purpose of this study is to obtain biologic materials from the blood, airways and/or urine of normal individuals and individuals with lung disease. The normal are used to establish a set of normal ranges for various parameters. These provide control information when compared to individuals with various pulmonary diseases, and will help in understanding of the etiology and pathogenesis of various lung diseases. The underlying hypothesis is that the pathologic morphological changes in the airway epithelium must be preceded by changes in the gene expression pattern of the airway epithelium and potentially in macrophages.

DETAILED DESCRIPTION:
This is a protocol to obtain blood, urine and/or airway specimens from normal individuals and individuals with lung disorders in order to carry out laboratory studies looking at genetic expression, gene transfer, infection, proteins, human genes, and to store specimens for future genetic studies. Specimens collected may include blood, urine and airway samples (nasal, airway brushing, biopsy and/or washings) from consenting subjects. Subjects will include both individuals diagnosed with lung disease and healthy control subjects. The purpose of this study is to obtain biologic materials from the blood, airways and/or urine of normal individuals and individuals with lung disease. The normal are used to establish a set of normal ranges for various parameters. These provide control information when compared to individuals with various pulmonary diseases, and will help in understanding of the etiology and pathogenesis of various lung diseases. The investigators will use bronchoscopy (inserting a scope into the lungs) to obtain airway cells by brushing, biopsy and/or washings in individuals with lung disease and in healthy controls. By studying those cells, the investigators hope to learn more about the specific causes of lung disease, how lung disease manifests and progresses, and how lung disease can be treated.

ELIGIBILITY:
Inclusion Criteria:

Group 1.1 - HEALTHY VOLUNTEER RESEARCH SUBJECTS (Healthy as defined by those not having lung disease and inclusive of: all races, ethnicities, sex, HIV status, smoking status and multiple birth status, etc., within the general population. Smoking status is defined for individuals that may use any of the following: cigarettes, pipes, E-cigarettes, waterpipe, shisha, etc.):

* All study subjects should be able to provide informed consent
* Males or females ages 18 years and older
* Must provide HIV informed consent

Group 1.2 - VOLUNTEER RESEARCH SUBJECTS WITH LUNG DISEASE (As defined by those having lung disease or symptoms of lung disease and inclusive of: all races, ethnicities, sex, HIV status, smoking status and multiple birth status, etc., within the general population. Smoking status is defined for individuals that may use any of the following: cigarettes, pipes, E-cigarettes, waterpipe, shisha, etc.):

* Must provide informed consent
* Males and females age 18 years and older
* Lung disease proven by at least one of the following: symptoms consistent with pulmonary disease; (2) chest X-rays consistent with lung disease; (3) pulmonary function tests consistent with lung disease; (4) lung biopsy consistent with lung disease; (5) family history of lung disease; and/or (6) diseases of organs with known association with lung disease
* Must provide HIV informed consent

Additional Inclusion criteria for CF subjects:

• All CF subjects will be homozygous for the ΔF508 mutation, with mild-moderate lung disease as defined by FEV1 ≥ 50%

Group 2 - WCMC/NYPH CLINICAL PATIENTS

* Must provide informed consent
* Males and females, age 18 years and older
* Lung disease proven by at least one of the following: (1) symptoms consistent with pulmonary disease; (2) chest X-rays consistent with lung disease; (3) pulmonary function tests consistent with lung disease; (4) lung biopsy consistent with lung disease; (5) family history of lung disease; (6) diseases of organs with known association with lung disease, and (7) individuals with the blood eosinophil levels of 5% or greater.

Group 3 - PCNY CLINICAL PATIENTS VOLUNTEER RESEARCH SUBJECTS WITH LUNG DISEASE

* Must provide informed consent
* Males and females, age 18 years and older
* Lung disease proven by at least one of the following: symptoms consistent with pulmonary disease; (2) chest X-rays consistent with lung disease; (3) pulmonary function tests consistent with lung disease; (4) lung biopsy consistent with lung disease; (5) family history of lung disease; and (6) diseases of organs with known association with lung disease

Exclusion Criteria:

Group 1.1 - HEALTHY VOLUNTEER RESEARCH SUBJECTS

* Individuals not deemed in good overall health by the investigator during screening visits and/or prior to the bronchoscopy will not be accepted into the study.
* Individuals with history of chronic lung disease, including asthma or with recurrent or recent (within three months) acute pulmonary disease will not be accepted into the study.
* Individuals with allergies to atropine or any local anesthetic will not be accepted into the study.
* Individuals with allergies to pilocarpine, isoproterenol, terbutaline, atropine or aminophylline will not be accepted into the study.
* Females who are pregnant or nursing will not be accepted into the study

Group 1.2 - VOLUNTEER RESEARCH SUBJECTS WITH LUNG DISEASE

* Any history of allergies to xylocaine, lidocaine, versed, valium, atropine, pilocarpine, isoproterenol, terbutaline, aminophylline, or any local anesthetic will not be included in the study
* Individuals deemed unable to complete the bronchoscopy due to health concerns by the investigator.
* Females who are pregnant or nursing

Additional Exclusion criteria for CF subjects:

* Experienced a recent (≤ 8 weeks) pulmonary exacerbation of their disease

Group 2 - WCMC/NYPH CLINICAL PATIENTS

* Patient refuses consent

Group 3 - PCNY CLINICAL PATIENTS

* Patient refuses consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: New York Metropolitan area residents
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2012-08-29 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Establishing normal ranges for various parameters | Participants upon completing the study will be followed up by a phone call seven days after their visit.
  The primary objective of the study is to obtain biologic materials from the blood, airways and/or urine of normal individuals and individuals with lung disease. The normal are used to establish a set of normal ranges for various parameters. These provide control information when compared to individuals with various pulmonary diseases, and will help in understanding the etiology and pathogenesis of various lung diseases.

SECONDARY OUTCOMES:
Learning about the genetic composition of the airway cells | Participants upon completing the study will be followed up by a phone call seven days after their visit.
  The secondary objective is to learn more about the genetic composition the cells that line the airways (windpipes) of the lungs in normal individuals and in individuals with lung disease.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G. Crystal, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College and Weill Cornell Medical Center, Department of Genetic Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Staudt MR, Salit J, Kaner RJ, Hollmann C, Crystal RG. Altered lung biology of healthy never smokers following acute inhalation of E-cigarettes. Respir Res. 2018 May 14;19(1):78. doi: 10.1186/s12931-018-0778-z. PMID 29754582
- [Derived] Strulovici-Barel Y, Staudt MR, Krause A, Gordon C, Tilley AE, Harvey BG, Kaner RJ, Hollmann C, Mezey JG, Bitter H, Pillai SG, Hilton H, Wolff G, Stevenson CS, Visvanathan S, Fine JS, Crystal RG. Persistence of circulating endothelial microparticles in COPD despite smoking cessation. Thorax. 2016 Dec;71(12):1137-1144. doi: 10.1136/thoraxjnl-2015-208274. Epub 2016 Jul 26. PMID 27462120